CLINICAL TRIAL: NCT02087137
Title: Functional Impact of a Memory Intervention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Susan Vandermorris, Ph.D., C.Psych., Psychologist, Baycrest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-21
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Aging
Keywords: aging; memory; memory training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memory and Aging Program (Active Comparator): The Memory and Aging Program intervention consists of five 2-hour sessions conducted over five consecutive weeks. The content of the program includes: (a) the provision of factual information (i.e., about memory, age-related memory changes, lifestyle factors affecting memory, and memory strategies) in an informal lecture format; and (b) memory intervention (i.e., practice and application of several evidence-based memory strategies) in a hands-on interactive format.
  Interventions: Behavioral: Memory and Aging Program
- Wait-list Control (No Intervention): Participants randomized to the wait-list control group will receive no intervention following randomization. They will be offered the intervention immediately following completion of the week 14 outcome testing session.

INTERVENTIONS:
Behavioral: Memory and Aging Program
  Arms: Memory and Aging Program

SUMMARY:
Normal aging is associated with decline in some aspects of memory, and this can be a risk factor for reductions in everyday functioning. The Baycrest Memory and Aging Program teaches positive adaptation to age-related memory changes, including strategies for minimizing the everyday impact of normal memory change and positive lifestyle change to maximize brain health. Prior research has shown that the Memory and Aging program is effective in increasing participants' knowledge about memory, use of memory strategies, and confidence in memory function, as well as adoption of healthier lifestyle practices and reduction in intention to use unneeded health care resources.

Although not one of the stated goals of the program, informal feedback from participants suggests that the educational content and skills training in the Memory and Aging Program has led some participants to change behaviours in ways that lead to significant improvements in their everyday functioning. For example, graduating participants often volunteer examples of how they have applied what they have learned to succeed in everyday memory tasks such as learning a new name or keeping track of future plans. Based on this participant feedback, it is hypothesized that the knowledge, skills, and confidence gained by Memory and Aging Program participants may lead to positive behaviour changes that, in turn, lead to improved everyday functioning. The present study will test this hypothesis using a randomized controlled pretest-posttest design.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-90
* Available to participate in all testing and intervention sessions (located in Toronto, Canada)

Exclusion Criteria:

* health conditions with major effects on cognition, including a current or previous history of stroke, brain surgery, or diagnosed neurological disorder
* dependence in instrumental activities of daily living
* cognitive impairment, defined as performance below cutoff for cognitive impairment on a standardized cognitive test, the Telephone Interview for Cognitive Status (Brandt, Spencer, & Folstein, 1988).
* affective impairment, defined as performance below cutoff for depression on standardized depression screen, the Geriatric Depression Scale (Yesavage et al., 1983)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in healthy lifestyle behaviours as measured by Health Promoting Lifestyle Profile II (Walker, Sechrist, & Pender, 1987) | Baseline, Week 8, week 14
Change from baseline in memory strategy use as measured by the Memory Strategy Toolbox (modified from Troyer, 2001) | Baseline, Week 8, week 14
Attainment of individualized goals for (a) lifestyle change, (b) memory strategy use, and (c) functional outcomes of memory strategy use as measured by Goal Attainment Scaling (Gordon, Powell, & Rockwood, 2000; Kiresuk, Smith, & Cardillo, 1994) | Baseline, Week 8, week 14

SECONDARY OUTCOMES:
Change in positive and negative affect as measured by Positive and Negative Affect Schedule (Watson, Clark, & Tellegen, 1988) | Baseline, Week 8, week 14
Change in general health status as measured by the RAND 36-Item Short-Form Health Survey (Ware & Sherbourne, 1992). | Baseline, Week 8, week 14
General Self-Efficacy Scale (Schwarzer & Jerusalem, 1995) | Baseline, Week 8, week 14
Prospective and Retrospective Memory Questionnaire (Smith, Della Sala, Logie, & Maylor, 2000) | Baseline, Week 8, week 14
Self-report health status, lifestyle changes, attitudes about aging | Baseline, Week 8, week 14

OTHER OUTCOMES:
Change in memory knowledge as measured by Memory knowledge quiz (modified from Troyer, 2001). | Baseline, Week 8, week 14
Change in self-perceived memory as measured by Multifactorial Metamemory Questionnaire (Troyer & Rich, 2002) | Baseline, 8 weeks, 14 weeks
Change in prospective memory function (Prospective telephone-call task, Troyer, 2001; actual week, Rendell & Craik, 2001) | Baseline, 8 weeks, 14 weeks
Change in name learning (Name-learning task, based on Troyer, Häfliger, Cadieux, & Craik, 2006) | Baseline, 8 weeks, 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan Vandermorris, PhD, Principal Investigator — Baycrest
Locations (1):
- Baycrest, Toronto, Ontario, Canada

REFERENCES:
- [Background] Brandt, J., Spencer, M., & Folstein, M. (1988). The Telephone Interview for Cognitive Status. Neuropsychiatry, Neuropsychology, & Behavioral Neurology, 1(2), 111-117.
- [Background] Gordon J, Rockwood K, Powell C. Assessing patients' views of clinical changes. JAMA. 2000 Apr 12;283(14):1824-5. No abstract available. PMID 10770141
- [Background] Kiresuk, T. J., Smith, A., & Cardillo, J. E. (1994). Goal attainment scaling: Applications, theory, and measurement. Hillsdale, NJ: Lawrence Erlbaum Associates.
- [Background] Troyer, A. K. (2001). Improving memory knowledge, satisfaction, and functioning via an education and intervention program for older adults. Aging, Neuropsychology, and Cognition, 8(4), 256-268.
- [Background] Troyer AK, Hafliger A, Cadieux MJ, Craik FI. Name and face learning in older adults: effects of level of processing, self-generation, and intention to learn. J Gerontol B Psychol Sci Soc Sci. 2006 Mar;61(2):P67-74. doi: 10.1093/geronb/61.2.p67. PMID 16497956
- [Background] Troyer AK, Rich JB. Psychometric properties of a new metamemory questionnaire for older adults. J Gerontol B Psychol Sci Soc Sci. 2002 Jan;57(1):P19-27. doi: 10.1093/geronb/57.1.p19. PMID 11773220
- [Background] Walker SN, Sechrist KR, Pender NJ. The Health-Promoting Lifestyle Profile: development and psychometric characteristics. Nurs Res. 1987 Mar-Apr;36(2):76-81. PMID 3644262
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Derived] Vandermorris S, Au A, Gardner S, Troyer AK. Initiation and maintenance of behaviour change to support memory and brain health in older adults: A randomized controlled trial. Neuropsychol Rehabil. 2022 May;32(4):611-628. doi: 10.1080/09602011.2020.1841656. Epub 2020 Nov 17. PMID 33203317
- [Derived] Herdman KA, Vandermorris S, Davidson S, Au A, Troyer AK. Comparable achievement of client-identified, self-rated goals in intervention and no-intervention groups: reevaluating the use of Goal Attainment Scaling as an outcome measure. Neuropsychol Rehabil. 2019 Dec;29(10):1600-1610. doi: 10.1080/09602011.2018.1432490. Epub 2018 Feb 12. PMID 29430998
- See also: Related Info — http://www.baycrest.org/memory